CLINICAL TRIAL: NCT06069960
Title: Sequential Adult Left Lateral Lobe Liver Transplantation (SALT) in Patients With Unresectable Colorectal Liver Metastases: a Single-center, Prospective, Single-arm Study
Brief Title: SALT for Unresectable Colorectal Liver Metastases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY2023-186-C
Record Dates: First submitted 2023-09-22; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Colon Cancer Liver Metastases
Keywords: liver transplantation; two-stage liver resection; colorectal liver metastases

STUDY DESIGN:
Intervention Model Description: SALT operation plan for patients who meet the enrollment conditions and successfully match the donor liver: Hemihepatectomy combined with left lateral lobe liver transplantation was performed first, and residual liver resection was performed after the graft grew to a sufficient functional liver volume.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical group (Experimental): SALT operation plan for patients who meet the enrollment conditions and successfully match the donor liver: Hemihepatectomy combined with left lateral lobe liver transplantation was performed first, and residual liver resection was performed after the graft grew to a sufficient functional liver volume.
  Interventions: Procedure: sequential adult left lateral lobe liver transplantation (SALT)

INTERVENTIONS:
Procedure: sequential adult left lateral lobe liver transplantation (SALT) — Hemihepatectomy combined with left lateral lobe liver transplantation was performed first, and residual liver resection was performed after the graft grew to a sufficient functional liver volume.

SUMMARY:
Colon cancer is a common malignancy with a low survival rate worldwide, and unresectable colon cancer liver metastases (ICRLM) have a worse prognosis. The liver is the most common metastatic organ of colorectal cancer, and palliative chemotherapy is the only option for most ICRLM patients. Regrettably, the median survival time of all patients receiving chemotherapy is only 2 years, and the 5-year survival rate is only 10%. Liver transplantation is an ideal choice for patients with ICRLM, which can significantly improve the postoperative survival rate. But the most serious problem facing such patients is the shortage of donor livers. In 2015, Norwegian scholars proposed a new surgical method, that is, resection and partial liver segment (2-3 segment) transplantation combined with delayed total hepatectomy can greatly alleviate the shortage of liver donors in the above-mentioned patients. Based on the experience of clinical operation, our center proposes and designs a clinical study of sequential adult left lateral lobe liver transplantation (SALT) for the treatment of iCRLM. On the basis of RAPID, the safety and efficacy of sequential adult left lateral lobe liver transplantation were evaluated for the above patients.

DETAILED DESCRIPTION:
Colorectal cancer is currently the third most common malignant tumor in the world, and about 20%-50% of patients have liver metastases at the time of diagnosis or progress to liver metastases thereafter. The liver is the most frequently invaded organ by colorectal cancer, and liver resection is considered to be the best and only treatment option for patients with colorectal liver metastases (CLMs). However, only about 20% of patients are candidates for radical hepatectomy. For most patients who are not candidates for hepatectomy, palliative chemotherapy is the only option. Regrettably, the median survival time of all patients receiving chemotherapy is only 2 years, and the 5-year survival rate is only 10%.

Theoretically, liver transplantation is an ideal choice for patients with unresectable colorectal liver metastases (Irresectable Colorectal Liver Metastases, iCRLM). In a clinical study in Norway, 21 patients with iCRLM were enrolled and treated with liver transplantation, although 19 patients had recurrence and metastasis after transplantation (median time 6 months, range 2-24 months). However, the 1-year, 3-year and 5-year survival rates rose to 95%, 68% and 60% after surgery. In this study, the risk factors for poor prognosis after liver transplantation in iCRLM patients were summarized: the largest tumor diameter was more than 5.5 cm, CEA before transplantation was >80ug/ml, the interval between primary disease surgery and transplantation was less than 2 years, and poor response to chemotherapy. Subsequently, the center conducted a second study and performed liver transplantation on 15 patients with iCRLM after optimizing the inclusion criteria. The 1-year, 3-year, and 5-year survival rates were 100%, 83%, and 83%, and the recurrence-free survival rates were 53%, 44%, and 35%. The above studies have proved that liver transplantation can significantly improve the prognosis of patients with iCRLM. However, the shortage of donor livers is the most serious problem faced by iCRLM patients. Moreover, iCRLM is generally considered a contraindication for liver transplantation, so it is more difficult for patients with iCRLM to obtain a donor liver.

Therefore, expanding the donor liver pool is urgently needed for the treatment of patients with iCRLM. In 2015, Norwegian scholars proposed a new surgical method, that is, resection and partial liver segment 2-3 transplantation with delayed total hepatectomy (RAPID) . This approach allows transplantation of the left liver (segments 2+3) to an adult recipient, while the remaining enlarged right hemi-liver is transplanted to another adult recipient, effectively avoiding some unsuitable left lateral lobe livers for pediatric recipients to be wasted. Recipients who received right-hemi-liver transplantation had a similar prognosis compared with those who received whole-liver transplantation. Therefore, if the RAPID technique is confirmed to be feasible, it can greatly alleviate the shortage of liver donors. In addition to cadaver sources, living adult donors can also be considered as the source of liver donors. A smaller left lateral lobe donor liver also places less burden on the donor than a left or right hemiliver.

To sum up, our center proposed and designed a clinical study of sequential adult left lateral lobe liver transplantation (SALT) in the treatment of patients with iCRLM based on clinical surgical experience. On the basis of RAPID surgery, the overall survival rate of patients with iCRLM was evaluated by SALT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75;
2. Physical fitness status (ECOG) 0~1;
3. Histologically confirmed primary colorectal neoplasm. The time from primary colorectal tumor resection to transplantation is ≥3 months and the stage of primary colorectal tumor is ≤T3N1. Accept T4N0 or T4N2 if primary tumor resection interval is ≥ 2 years
4. Liver metastases (CRLM) located in bilateral livers, or limited to liver and unresectable CRLM after discussion by MDT;
5. According to PET/CT, CT and MRI, there are no other abdominal metastases except the liver or 1-3 resectable lung metastases;
6. Patients have received at least 6-8 weeks of first-line chemotherapy at the time of screening. According to RECIST criteria, CRLM was stable or partially regressed during and after treatment (still not completely resectable);
7. The CEA (carcinoembryonic antigen) value before screening is ≤80 µg/L or the highest level after treatment is reduced by ≥ 50%;
8. Sign the informed consent form.

Exclusion Criteria:

1. Extrahepatic tumor burden (except for resectable lung metastases) and/or large vessel tumor infiltration;
2. The largest liver tumor lesion >5.5cm at the time of screening;
3. Tumor progression during chemotherapy or severe comorbidities that make transplantation impossible;
4. BRAF mutation and/or microsatellite instability primary tumor (MSI);
5. Suffering from other primary malignant tumors in the past 5 years;
6. Cardiopulmonary disease that cannot be corrected, with high surgical risk, or anatomical abnormality that makes liver transplantation impossible;
7. Substance abuse, medical, psychological or social conditions may interfere with the patient's participation in the study or evaluation of the study results;
8. Combined with AIDS and other diseases that affect surgery or tumor progression;
9. Pregnant or lactating patients;
10. Other reasons that the researchers think are not suitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival（OS） | 3 years after the second liver resection
  To describe overall survival in patients with unresectable colorectal cancer liver metastases treated with sequential adult left lateral lobe liver transplantation.

SECONDARY OUTCOMES:
Disease-free survival，DFS | 1 month, 3 months, 6 months, 1 year, 2 years and 3 years post-transplant
  Describe the tumor-free survival period of SALT in the treatment of iCRLM

IPD SHARING:
Plan to Share IPD: No